CLINICAL TRIAL: NCT05616078
Title: Laser Versus Cryotherapy for the Treatment of Recalcitrant Warts: a Randomised Controlled Trial
Brief Title: Laser Versus Cryotherapy for the Treatment of Recalcitrant Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The 306 Hospital of People's Liberation Army (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 306PLA-004
Record Dates: First submitted 2022-11-01; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Warts
MeSH Terms: conditions — Warts | interventions — Laser Therapy; Cryotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser treatment (Experimental): LP-Nd:YAG laser treatment
  Interventions: Other: laser treatment
- cryotherapy (Active Comparator): cryotherapy with liquid nitrogen
  Interventions: Other: cryotherapy

INTERVENTIONS:
Other: laser treatment — a maximum of 4 sessions, with an interval of 3 to 4 weeks
  Arms: laser treatment
Other: cryotherapy — a maximum of 4 sessions, with an interval of 3 to 4 weeks
  Arms: cryotherapy

SUMMARY:
To evaluate whether laser was superior to cryotherapy for recalcitrant warts

DETAILED DESCRIPTION:
Patients with recalcitrant warts were randomized equally to receive laser or cryotherapy every 3 to 4 weeks, for a maximum of 4 sessions.The primary outcomes were the cure rate at 16 weeks; secondary outcomes included time to clearance of warts, patient satisfaction with the treatment and treatment-related adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HPV2/27/57-induced recalcitrant warts, including periungualor mosaic warts, common or plantar warts with a duration of longer than 1 year, and common or plantar warts previously received no more than two sessions of cryotherapy
* Total number of warts is ≤10 .
* Aged 18 years or older.

Exclusion Criteria:

* Patients are currently participating in another trial for the treatment of cutaneous warts.
* Patients have taken immunosuppressant drugs (such as oral corticosteroids) during the past three months.
* Patients have impaired healing eg due to diabetes, vitamin A deficiency, hyperthyroidism and hypothyroidism.
* Patients have autoimmune diseases (such as systemic lupus erythematosus, dermatomyositis, scleroderma or other diseases).
* Patients are pregnant or ready for pregnancies or breast-feeding.
* Patients have cold intolerance (such as cold urticaria, cryoglobulinaemia, cold agglutinin syndrome or Raynaud's syndrome).
* Patients have local pain intolerance.
* Patients have local hypoesthesia.
* Patients are unable to tolerate laser or cryotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
cure rate at 16 weeks | 16 weeks since the initial treatment
  A patient was considered to be cured if all warts were no longer visible and could not be palpated anymore.

SECONDARY OUTCOMES:
time to clearance of warts | 16 weeks since the initial treatment
  The time from treatment initiation until clearance of all warts
patient satisfaction with the treatment | 16 weeks since the initial treatment
  Patient satisfaction was rated on a 5-point scale (from very happy to very unhappy)
treatment-related adverse events | 16 weeks since the initial treatment
  Some adverse effects, including pain, swelling, blisters, hemorrhagic bullae, bruising, and skin breakdown, were recorded by the patients, whereas others, including secondary bacterial infection, hyperpigmentation, hypopigmentation, and scarring were evaluated by a dermatologist

CONTACTS AND LOCATIONS:
Overall Officials: Shichao Lu, MD, Principal Investigator — The 306 Hospital of People's Liberation Army